CLINICAL TRIAL: NCT01838096
Title: Alumina Matrix Composite Ceramic Bearing Total Hip Arthroplasty in Patients Younger Than 30 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: CeramTec GmbH (Unknown)
Responsible Party: Principal Investigator, Kyung-Hoi Koo, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cera-001
Record Dates: First submitted 2013-04-15; First posted 2013-04-23 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Advanced Hip Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- THA (Experimental)
  Interventions: Device: THA using 4th generation CoC

INTERVENTIONS:
Device: THA using 4th generation CoC

SUMMARY:
This study will evaluate clinical outcome on patients who undergo cementless 4th generation ceramic (BIOLOX®delta, CeramTec GmbH, Plochingen, Germany) on ceramic (CoC) bearing total hip aArthroplasty ("THA") in patients younger than 30 years.

ELIGIBILITY:
Inclusion Criteria:

* younger than 30 years
* advanced hip disease

Exclusion Criteria:

* older than 30 years

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2008-03; Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
survival rate of 4th generation ceramic-on-ceramic THA | 5 years
  survival rate of 4th generation ceramic-on-ceramic THA end point for best senario ; any reoperation end point for moderate senario ; loosening end point for worst senario ; osteolysis

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Hoi Koo, Professor, Principal Investigator — Seoul National University Bundang Hospital

REFERENCES:
- [Derived] Lee YK, Kim KC, Yoon BH, Kim TY, Ha YC, Koo KH. Cementless total hip arthroplasty with delta-on-delta ceramic bearing in patients younger than 30 years. Hip Int. 2021 Mar;31(2):181-185. doi: 10.1177/1120700019889592. Epub 2019 Nov 25. PMID 31766869